CLINICAL TRIAL: NCT07036445
Title: Comparison of Interlaminar CT Guided Epidural Platelet Rich Plasma Versus Steroid Injection in Patients With Lumbar Radicular Pain : a Prospective Study With Long Term Follow up
Brief Title: Comparison of Interlaminar CT Guided Epidural Platelet Rich Plasma Versus Steroid Injection in Patients With Lumbar Radicular Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique du Sport, Bordeaux Mérignac (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-38-SBM
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Herniated Disc
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- steroid treatment (Active Comparator)
  Interventions: Procedure: Epidural Steroid Injection
- platelet-rich plasma treatment (Experimental)
  Interventions: Procedure: Epidural platelet-rich plasma injection

INTERVENTIONS:
Procedure: Epidural Steroid Injection — Intervention consists of interlaminar CT guided epidural steroid injection
  Arms: steroid treatment
Procedure: Epidural platelet-rich plasma injection — Intervention consists of interlaminar CT guided epidural platelet-rich plasma injection after recovery of plasma by blood sampling and centrifugation
  Arms: platelet-rich plasma treatment

SUMMARY:
The treatment of persistent lumbar radicular pain (LRP) using CT-guided epidural steroid injection (ESI) is widely used and associated with rare but serious complications. Platelet-rich plasma (PRP), which has recently been shown to promote healing and the anti-inflammatory process by delivering growth factors and cytokines, could be an alternative and potentially safer option. A previous study showed that PRP was as effective as ESI in treating this condition, without major complications.

This study aims to compare these two treatments over the long term (2 years).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral resistant LRP associated with a herniated disc on MRI images. (Diagnosis of resistance after 6 weeks of appropriate medical treatment).

Exclusion Criteria:

* Patients with infections,
* Patients who have had previous percutaneous corticosteroid injections,
* Patients undergoing systemic corticosteroid treatment,
* Patients with immune deficiencies,
* Patients who are allergic to the contrast medium used,
* Pregnant or breastfeeding patients,
* Patients with a history of allergies to anesthetics or corticosteroids,
* Anticoagulant treatment or blood disorders, patients on antiplatelet therapy
* Taking NSAIDs within two weeks prior to the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional ability | 30 minutes before procedure ; 6 weeks after procedure ; 6 months, 1 year, 2 years after procedure
  Oswestry Disability Questionnaire ranging from 0 to 100%

SECONDARY OUTCOMES:
Pain evaluation | 6 weeks, 6 months, 1 year and 2 years after procedure
  Numerical pain rating scale (NRS): intensity of combined pain in the legs and back ranging from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du Sport, Mérignac, France

IPD SHARING:
Plan to Share IPD: No